CLINICAL TRIAL: NCT02217501
Title: Antiplatelet Strategy for Peripheral Arterial Interventions for Revascularization of Lower Extremities
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Subhash Banerjee, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 122013-065; NCT02317822 (obsolete NCT alias)
Record Dates: First submitted 2014-08-01; First posted 2014-08-15 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease, antiplatelet therapy
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAPT - clinically indicated duration+12m (Experimental): Clopidogrel 75 mg daily and Acetylsalicylic acid (ASA) 75-100 mg daily for clinically indicated duration plus an additional 12 months
  Interventions: Drug: Clopidogrel; Drug: Acetylsalicylic acid (ASA)
- DAPT - clinically indicated duration (Active Comparator): Clopidogrel 75 mg daily and Acetylsalicylic acid (ASA) 75-100 mg daily for clinically indicated duration with a minimum of 30 days
  Interventions: Drug: Clopidogrel; Drug: Acetylsalicylic acid (ASA)

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg once daily for clinically indicated duration or for clinically indication duration + 12 months
  Other Names: Plavix
Drug: Acetylsalicylic acid (ASA) — Acetylsalicylic acid (ASA) 75-100 mg once daily for clinically indicated duration or for clinically indication duration + 12 months
  Other Names: Aspirin

SUMMARY:
The purpose of this study is to evaluate whether clopidogrel 75 mg daily on a background of aspirin 75-100 mg/d for clinically indicated duration or for an additional 12 months will lead to an increased rate of primary patency, limb salvage, non-fatal myocardial infarction (MI), ischemic stroke, and survival, in patients receiving endovascular treatment of PAD at end of study treatment.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is extremely prevalent worldwide and affects over 206 million people. Over 36 million patients with PAD are estimated to be present in the United States. Percutaneous revascularization therapies have evolved dramatically, yet the long-term success of these therapies remains modest and the morbidity and mortality associated with PAD remains high, with up to 30% mortality risk at 5 years. Nearly, 3.2 million endovascular procedures are performed annually. Though, this exceeds interventional procedures performed for coronary artery disease (CAD), the current PAD guidelines are silent regarding the need and optimal duration of antiplatelet therapy (APT) for patients following an endovascular procedure for claudication or critical limb ischemia (CLI). The lack of data and clinical studies is by far the greatest impediment to the formulation of such guideline recommendations critically needed by providers and patients alike, especially given the current limited durability of lower extremity endovascular procedures.

The objective of this trial is to evaluate whether clopidogrel 75 mg QD on a background of ASA 75-100 mg/d for clinically indicated duration or for an additional 12 months will lead to an increased rate of primary patency, limb salvage, non-fatal myocardial infarction (MI), ischemic stroke, and survival, in patients receiving endovascular treatment of PAD at end of study treatment.

The investigators hypothesize that dual antiplatelet therapy (DAPT) with ASA and clopidogrel administered for an additional 12 months following iliac, femoropopliteal or below the knee endovascular intervention will improve primary patency, limb salvage, freedom from ischemic stroke and survival, in patients with symptomatic PAD.

Clinical endpoints will be analyzed in all subjects who are enrolled, regardless of whether the trial treatment administered successfully completed for the desired duration. A subject will be considered enrolled in the trial when he/she is randomized to one of the treatment arms of the study. All endpoints are subject-based unless otherwise specified.

The primary endpoint is subject-based of the longer of a 12-month or end of study treatment endpoint of the first occurrence of index limb arterial occlusion, surgical intervention, endovascular intervention, amputation of the affected limb (primary patency and limb salvage), MI, ischemic stroke or death (survival).

The secondary endpoints are subject-based on the longer of a 12 month or end of study treatment endpoints that include: (a) the first occurrence of any individual component of the primary endpoint, (b) the first occurrence of the following during follow-up: cardiovascular death, or MI, or ischemic stroke, or any amputation above the ankle and (c) severe bleeding defined according to the Global Utilization of Streptokinase and Tissue plasminogen activator for Occluded coronary arteries (GUSTO) classification.

The tertiary endpoint is based on the longer of a 12-month or end of study moderate bleeding according to the GUSTO classification.

ELIGIBILITY:
Inclusion Criteria:

General:

* Signed informed consent
* At least 18 years old
* Documented symptomatic iliac, femoropopliteal (FP) or below-the knee artery (BTK) atherosclerotic disease (Rutherford/Becker category 2, 3 or ≥4)
* Undergone clinically indicated uncomplicated endovascular intervention to one or more locations of the iliac, femoropopliteal below-the knee arteries
* Estimated survival ≥1 year in the judgment of the primary operator
* Pre-index procedure use of ASA, clopidogrel or both at any dose

Angiographic:

* De novo or restenotic lesions in the common and/or external iliac artery, superficial femoral artery (SFA), popliteal artery, tibio-peroneal (TP) trunk, anterior tibial (AT) artery, peroneal artery (PA) or posterior tibial (PT) artery (applies to all target lesions if multiple)
* Subjects with multiple planned procedures can be enrolled after the completion of the last planned procedure.

Exclusion Criteria:

General:

* Complicated qualifying procedure (perforation, flow limiting dissection, distal embolization requiring re-intervention, need for repeat endovascular, surgical revascularization, amputation or blood transfusion prior to hospital discharge following an index procedure
* Extended hospital stay >7 days following the index procedure
* Allergy to aspirin or clopidogrel
* Life expectancy less than 12 months due to other medical co-morbid condition(s) that could limit the subject's ability to participate in the trial, limit the subject's compliance with the follow-up requirements, or impact the scientific integrity of the trial
* Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated.
* Intolerance to antiplatelet, anticoagulant, or thrombolytic medications
* Platelet count <90,000 mm3 or >600,000 mm3
* Serum creatinine >2.5 mg/dL
* Dialysis-dependent end stage renal disease
* Pregnancy
* Current participation in another drug or device trial that requires interruption of dual-antiplatelet therapy with aspirin or clopidogrel for the duration of the study
* Planned surgeries, endovascular or other non-vascular or cardiac procedures
* Concurrent warfarin or other chronic oral anticoagulant therapy
* Contraindication(s) to the use of AT (history of intra-cerebral bleed, presence of intra-cerebral mass, recent or <6 weeks gastrointestinal bleed, blood transfusion within the last 6 weeks, any trauma requiring surgery or blood transfusion within the last 4 weeks or any surgical procedure within the last 4 weeks.

Angiographic:

* Endovascular intervention to iliac, femoropopliteal or BTK artery bypass graft
* Persistent, intraluminal thrombus of the proposed target lesion at the completion of the index procedure
* Perforated vessel as evidenced by extravasation of contrast media
* Vascular graft, aneurysm or postsurgical stenosis of the target vessel

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-11; Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — University of Texas Southwestern Medical Center; Subhash Banerjee, MD, Study Chair — University of Texas Southwestern Medical Center
Locations (4):
- United States (4):
  - Denver VA Medical Center, Denver, Colorado
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - VA North Texas Health Care System, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study results will be posted on clinical.trials.gov and through publications and presentations

REFERENCES:
- [Background] Hirsch AT, Duval S. The global pandemic of peripheral artery disease. Lancet. 2013 Oct 19;382(9901):1312-4. doi: 10.1016/S0140-6736(13)61576-7. Epub 2013 Aug 1. No abstract available. PMID 23915884
- [Background] Parikh SV, Saya S, Divanji P, Banerjee S, Selzer F, Abbott JD, Naidu SS, Wilensky RL, Faxon DP, Jacobs AK, Holper EM. Risk of death and myocardial infarction in patients with peripheral arterial disease undergoing percutaneous coronary intervention (from the National Heart, Lung and Blood Institute Dynamic Registry). Am J Cardiol. 2011 Apr 1;107(7):959-64. doi: 10.1016/j.amjcard.2010.11.019. Epub 2011 Jan 20. PMID 21256469
- [Background] Diehm C, Schuster A, Allenberg JR, Darius H, Haberl R, Lange S, Pittrow D, von Stritzky B, Tepohl G, Trampisch HJ. High prevalence of peripheral arterial disease and co-morbidity in 6880 primary care patients: cross-sectional study. Atherosclerosis. 2004 Jan;172(1):95-105. doi: 10.1016/s0021-9150(03)00204-1. PMID 14709362
- [Background] Hankey GJ, Norman PE, Eikelboom JW. Medical treatment of peripheral arterial disease. JAMA. 2006 Feb 1;295(5):547-53. doi: 10.1001/jama.295.5.547. PMID 16449620
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery/Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines. ACC/AHA Guidelines for the Management of Patients with Peripheral Arterial Disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Associations for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (writing committee to develop guidelines for the management of patients with peripheral arterial disease)--summary of recommendations. J Vasc Interv Radiol. 2006 Sep;17(9):1383-97; quiz 1398. doi: 10.1097/01.RVI.0000240426.53079.46. No abstract available. PMID 16990459
- [Background] Banerjee S, Das TS, Abu-Fadel MS, Dippel EJ, Shammas NW, Tran DL, Zankar A, Varghese C, Kelly KC, Weideman RA, Little BB, Reilly RF, Addo T, Brilakis ES. Pilot trial of cryoplasty or conventional balloon post-dilation of nitinol stents for revascularization of peripheral arterial segments: the COBRA trial. J Am Coll Cardiol. 2012 Oct 9;60(15):1352-9. doi: 10.1016/j.jacc.2012.05.042. Epub 2012 Sep 12. PMID 22981558
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646

RESULTS

PARTICIPANT FLOW:
Groups:
- DAPT - Clinically Indicated Duration: Clopidogrel 75 mg daily and Acetylsalicylic acid (ASA) 75-100 mg daily for clinically indicated duration with a minimum of 30 days
  Clopidogrel: Clopidogrel 75 mg once daily for clinically indicated duration or for clinically indication duration
  Acetylsalicylic acid (ASA): Acetylsalicylic acid (ASA) 75-100 mg once daily for clinically indicated duration or for clinically indication duration
Period: Overall Study
Arm/Group | DAPT - Clinically Indicated Duration+12m | DAPT - Clinically Indicated Duration
Started | 77 | 82
Completed | 74 | 78
Not Completed | 3 | 4
Not completed — Death | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DAPT - Clinically Indicated Duration+12m | DAPT - Clinically Indicated Duration | Total
Number analyzed (Participants) | 77 | 82 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.62 (8.82) | 65.27 (8.90) | 65.44 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 65 | 68 | 133
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Target Vessel Occlusion, Surgical Revascularization, Endovascular Revascularization, Major Amputation of Target Limb, Ischemic Stroke, MI, or Death
Description: Occlusion of the target vessel documented by any imaging procedure (eg, Duplex ultrasonography scan including B mode imaging and Doppler ultrasound scan) at any follow-up visit within 12 months or end of study treatment period, whichever is longer.
Time Frame: 12 months from index procedure or end of study treatment, whichever is longer, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | DAPT - Clinically Indicated Duration+12m | DAPT - Clinically Indicated Duration
Number analyzed (Participants) | 77 | 82
Participants | 13 | 16

2. Secondary Outcome: Number of Participants With First Occurrence of Bleeding
Description: Any mild, moderate, severe, or life-threatening bleeding.
  Severe or Life-threatening: Intracerebral hemorrhage Resulting in substantial hemodynamic compromise requiring treatment Moderate: Requiring blood transfusion but not resulting in hemodynamic compromise Mild: Bleeding that does not meet above criteria
  Severe bleeding defined according to the Global Utilization of Streptokinase and Tissue plasminogen activator for Occluded coronary arteries (GUSTO) classification.
Time Frame: 12 months from index procedure or end of study treatment, whichever is longer, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | DAPT - Clinically Indicated Duration+12m | DAPT - Clinically Indicated Duration
Number analyzed (Participants) | 77 | 82
Participants | 5 | 4
Statistical Analysis 1: Comparison: DAPT - Clinically Indicated Duration+12m vs DAPT - Clinically Indicated Duration; Test type: Superiority; p = 0.6595, Cochran-Mantel-Haenszel — Alpha of 0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time on informed consent and up to 18 months.
Arm/Group | DAPT - Clinically Indicated Duration+12m | DAPT - Clinically Indicated Duration
All-Cause Mortality (participants affected / at risk) | 3/77 | 4/82
Serious Adverse Events (participants affected / at risk) | 27/77 | 37/82
Other Adverse Events (participants affected / at risk) | 1/77 | 1/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPT - Clinically Indicated Duration+12m (N=77) | DAPT - Clinically Indicated Duration (N=82)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 3 (3)
Stroke (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Repeat Endovascular Revascularization (Vascular disorders) | 13 (13) | 16 (16)
Amputation (Surgical and medical procedures) | 7 (7) | 12 (12) — Amputation (major and minor)
Bleeding (Blood and lymphatic system disorders) | 3 (3) | 2 (2) — Bleeding required to be hospitalized.
Bleeding requiring transfusion (Surgical and medical procedures) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPT - Clinically Indicated Duration+12m (N=77) | DAPT - Clinically Indicated Duration (N=82)
CT/MR Angiography (Surgical and medical procedures) | 1 (1) | 1 (1) — CT/ MR Angiography

LIMITATIONS AND CAVEATS:
Study was not able to reach the target number of participants needed to achieve target power and statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT02217501/Prot_SAP_000.pdf